CLINICAL TRIAL: NCT02522741
Title: Safe Mothers, Safe Children Initiative
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 11-00175
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Child Maltreatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Parenting STAIR (Experimental)
  Interventions: Behavioral: Parenting STAIR

INTERVENTIONS:
Behavioral: Parenting STAIR — Parenting-STAIR is an adaptation of a 16 session study therapy entitled Skills Training in Affective and Interpersonal Regulation/Modified Prolonged Exposure (STAIR/MPE). It generally is comprised of approximately 23 sessions and includes seven didactic interaction parenting sessions. There are threskill building in areas such as e modules within Parenting STAIR: 1) Module 1 focuses on skill building (awareness of emotional states, management of negative feelings, regulation of emotional intensity, etc.); 2) Module 2 involves the processing of memories of trauma and creating a coherent and meaningful life narrative; 3) Module 3 includes both the mother and child, and focuses on increasing maternal attunement and improving parenting skills.

SUMMARY:
The purpose of this study is to evaluate the efficacy of an evidence-based post-traumatic stress disorder (PTSD) intervention adapted to focus on parenting-related impairment for mothers receiving preventive services. The study intervention is adapted from Skills Training in Affective and Interpersonal Regulation (STAIR). The investigators expect that the adaption (Parenting STAIR) has the potential to prevent child maltreatment as well as improve maternal and child well-being by reducing the effects of maternal PTSD and depression on parenting.

The investigators plan to recruit mothers with high levels of trauma-related symptoms from preventive service agencies, and invite them to participate in the study. This study is a single group design, and data will be collected pre-treatment, post-treatment, and 12-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who are receiving preventive services at the time of study enrollment and have histories of trauma, have symptoms of PTSD, without a history of psychotic disorder, or current domestic violence or substance abuse
* Have a child within the 2-9 age range, and are the child's primary caretaker
* Can communicate in English and/or Spanish

Exclusion Criteria:

* Women who have a history of psychotic disorder and/or who meet current DSM-IV criteria for abuse of drug or alcohol
* Women who are experiencing domestic violence at the time of the assessment
* Pregnant women are excluded from this pilot study because they are a potentially particularly vulnerable population. However, women who become pregnant while participating in the study will not be excluded
* Women who report suicidal ideation in the past two weeks on the SCID, or have a history of a suicide attempt during the last year as reported during the SCID interview
* Children who meet diagnostic criteria for developmental disorders (e.g., autism and mental retardation), and/or have a history of childhood psychosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The Clinician Administered PTSD Scale | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
Posttraumatic Stress Diagnostic Scale | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
Center for Epidemiological Studies Depression Scale | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
The Structured Clinical Interview for the Diagnostic & Statistical Manual of Mental Disorders (DSM)-IV Axis I Disorders | At baseline
Woman Abuse Screening Tool | At baseline
Strengths and Difficulties Questionnaire | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
Eyberg Child Behavior Inventory | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
Developmental Questionnaire | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
Traumatic Events Screening Inventory - Parent Report Revised, Trauma Symptom Checklist for Young | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)

SECONDARY OUTCOMES:
The Parenting Stress Index-Short Form | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
The Conflict Tactics Scale-Parent-Child | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
The Adult-Adolescent Parenting Inventory-2 | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
CAGE Substance Abuse Screening Tool | At baseline for individuals not meeting criteria for PTSD
Yale University PRIME Screening Test | At baseline for individuals not meeting criteria for PTSD
Connor-Davidson Resilience Scale | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
Interpersonal Support Evaluation List | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
Life Orientation Test-Revised | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
State Trait Anger Expression Inventory-2 | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
Difficulties of Emotional Regulation Scale | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)
Treatment Services Review | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatme
Working Alliance Inventory Short Form for Clients | Change from baseline to end of treatment (approximately 23 sessions over 23 weeks); change to post-treatment (12 weeks after completion of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Claude Chemtob, Principal Investigator — NYU MEDICAL CENTER
Locations (1):
- NYU Langone Medical Center, New York, New York, United States